CLINICAL TRIAL: NCT04029441
Title: he Effact of Helicobacter Hylori Eradication on the Development of Gastric Mucosa Pathology
Brief Title: The Effact of Helicobacter Hylori Eradication on the Development of Gastric Mucosa Pathology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Other Study IDs: 2018SDU-QILU-G115
Record Dates: First submitted 2019-07-21; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Helicobacter Gastritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — gastric mucosa
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the successful eradication cohort: the subjects who eradicate the Hp successfully after recieving the therapy or rescue therapy based on antimicrobial susceptibility test
  Interventions: Other: the eradication Hp
- the failure eradication cohort: the subjects who fail to eradicate the Hp after recieving the therapy or rescue therapy based on antimicrobial susceptibility test

INTERVENTIONS:
Other: the eradication Hp — the eradication of Hp based on antimicrobial susceptibility test
  Groups: the successful eradication cohort

SUMMARY:
Subjects who are included will recieve Hp eradication therapy based on antimicrobial susceptibility test. After the therapy, the subjects will be divided into two groups, the successful group and the failure group. And then they wiil be followed up to observe the development of the gastric mucosa pathology.

DETAILED DESCRIPTION:
Subjects who are included will recieve Hp eradication therapy based on antimicrobial susceptibility test. After the therapy, the subjects will be divided into two groups, the successful group and the failure group. The subjects who fail to eradicate the Hp after initial treatment and rescue treatment will go into the failure group. Otherwhile, they will go to the successful group.And then they wiil be followed up to observe the development of the gastric mucosa pathology. For mild atrophy gastritis, non- intestinal metaplasial gastritis, follow-up is performed every 2-3 years.For severe atrophy gastritis, intestinal metaplasial gastritis, follow-up is performed every 1-2 years. For patients wth high-grade intraepithelial neoplasia, they can be included 3 months after the endoscopic treatment, and the follow up will be performed at 6, 12 months after the treatment and then the follow up will be carried out every 1 year. For non-atrophic gastritis, no follow-up will be performed. All included patients will recieve a follow-up at the endpoint of 5 years. The follow-up includes endoscopy examination and serum test of PG I,PG II and gastrin 17.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged between 18 and 70 years old, with positive H. pylori infection that was not eradicated by previous therapies are included. The H. pylori infection is confirmed by the positive rapid urease test or 13C-breath test.

Exclusion Criteria:

* Patients with significant underlying disease including liver, cardiac, pulmonary, and renal diseases, neoplasia, coagulopathy and genetic diseases, history of gastric surgery, pregnancy, breast-feeding, active gastrointestinal bleeding, patients with peptic ulcer, the use of PPI, NSAID or antibiotics during the 4 weeks prior to enrolment, and previous history of allergic reactions to any of the medications used in this protocol. Patients previously treated with H. pylori eradication regimens or those unwilling to participate in the study were also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, aged between 18 and 70 years old, with positive H. pylori infection that was not eradicated by previous therapies are included.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
the pathologic status of mucosa | 5 years
  the development or change pathologic status of mucosa

SECONDARY OUTCOMES:
PG I | 5 years
  the serum level of PG I
PG II | 5 years
  the serum level of PG II
gastrin 17 | 5 years
  the serum level of gastrin 17

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli H Zuo, Study Chair — Qilu Hospital of Shandong University; Tian H Ma, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hosipital, Jinan, Shandong, China